CLINICAL TRIAL: NCT06367764
Title: LGBTQIA+ Initiative for Empowerment, Support, Coping, and PTSD Education: A Comparative Effectiveness Study of PTSD Treatments Among Sexual and Gender Minority Populations
Brief Title: A Comparative Effectiveness Study of PTSD Treatments Among Sexual and Gender Minority Populations
Acronym: LIFESCAPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Annesa Flentje, Professor of Medicine (Stanford Prevention Research Center), Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 79658; P0566840 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: PTSD
Keywords: PTSD; Therapy; LGBTQ; Depression; Comparative Effectiveness Trial; Substance Use; Minority Stress
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Processing Therapy (Active Comparator): Cognitive Processing Therapy is a ~12 session trauma-focused therapy that teaches cognitive restructuring skills to help clients change beliefs and process emotions related to a specific traumatic event, which can be generalized to other traumatic experiences as well as everyday stressors. After initial psychoeducation and practice with cognitive restructuring skills, patients use skills to identify and challenge maladaptive beliefs about the traumatic event itself as well as those related to five themes thought to be affected by trauma-safety, trust, power, control, esteem, and intimacy.
  Interventions: Behavioral: Cognitive Processing Therapy
- STAIR Narrative Therapy (Active Comparator): STAIR Narrative Therapy is a ~16-session multicomponent therapy that includes a coping skills component (10 sessions) focused on increasing skills in emotion regulation and interpersonal relationships to address day-to-day life stressors and improve functioning, and a trauma-focused component (6 sessions) which reviews a patient-selected series of traumatic experiences in which the meaning of the events is re-appraised particularly regarding sense of self and relationship to others.
  Interventions: Behavioral: STAIR Narrative Therapy

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy — Cognitive Processing Therapy teaches cognitive restructuring skills to help clients change beliefs and process emotions related to a traumatic event or events.
  Arms: Cognitive Processing Therapy
Behavioral: STAIR Narrative Therapy — STAIR Narrative Therapy teaches coping skills (e.g., for emotional regulation, interpersonal relationships, everyday stress) and includes a narrative trauma-focused component.
  Arms: STAIR Narrative Therapy

SUMMARY:
The goal of this clinical trial is see if Cognitive Processing Therapy and STAIR Narrative Therapy work to treat posttraumatic stress disorder (PTSD) among lesbian, gay, bisexual, transgender, queer/questioning, intersex, asexual/aromantic, and all other sexual or gender minority (LGBTQIA+) adults. The main questions it aims to answer are:

* Do these treatments reduce PTSD symptoms in LGBTQIA+ patients?
* Do these treatments help improve quality of life and reduce depression in LGBTQIA+ patients?
* Do stress from stigma and discrimination and drug/alcohol use change the impact of the treatment on PTSD symptoms?
* Are LGBTQIA+ patients satisfied with these treatments? Do these treatments work differently among different groups within the LGBTQIA+ community?
* Do LGBTQIA+ patients complete these treatments?

Study participants will receive one of these two PTSD treatments. Participants will complete assessments before and after receiving treatment.

DETAILED DESCRIPTION:
This study will compare two PTSD treatments that are known to work: Cognitive Processing Therapy (CPT) and STAIR Narrative Therapy (SNT). PTSD treatments have not been tested among LGBTQIA+ people. The study is trying to learn which treatment(s) work the best for LGBTQIA+ people in real world settings. This study will help guide clinical decision-making and the selection of PTSD treatment by health care organizations, clinicians, and patients based on what works best for LGBTQIA+ people.

The study will investigate which treatments work better in reducing PTSD symptoms among LGBTQIA+ people. The study will identify if minority stress (e.g., experiences of stigma and discrimination) and use of drugs or alcohol will moderate the effects of the interventions on PTSD symptoms. This study is investigating if both treatments improve depression symptoms and improve quality of life, and which treatments patients complete. The study is also examining if these treatments are effective for all individuals in the study, and if the effects of treatment are different among: 1) cisgender sexual minority men, cisgender sexual minority women, gender expansive or non-binary individuals, transgender women, transgender men, 2) participants who live in urban versus rural or suburban areas, and 3) racial and ethnic minority LGBTQIA+ participants.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Currently live in California
3. Ability to understand study procedures and to comply with them for the entire length of the study
4. Ability to understand a written informed consent document and the willing to sign it
5. Ability to speak and read English or Spanish
6. Identify as a sexual and/or gender minority
7. Score 33 or higher on the PTSD Checklist-5 (PCL-5)
8. Interest in getting treatment for PTSD
9. Not be in another concurrent psychotherapy treatment (group or individual) for PTSD (psychotherapy treatment for non-PTSD conditions is allowed).
10. Able to attend treatment sessions in person in San Francisco or have access to a device that allows for treatment via videoconferencing.

Exclusion Criteria:

1. Contraindication to any study-related procedure or assessment
2. Clinically significant impairment which interferes with ability to fully participate in the study (including symptoms of schizophrenia, schizoaffective disorder, bipolar disorder, or other disorders)
3. Active suicidal intent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Change in Posttraumatic Stress Disorder (PTSD) Symptoms Measured by PTSD Checklist for DSM-5 (PCL-5) | Months 0 (baseline), 3, 6, and 12
  The PCL-5 is a validated measure of self-report DSM-5 symptoms of PTSD. The self-report rating scale is 0-4 for each symptom, with higher scores indicating greater symptom severity.

SECONDARY OUTCOMES:
Change in Depression Measured by Patient Health Questionnaire (PHQ-9) | Months 0 (baseline), 3, 6, and 12
  The PHQ-9 is a 9-item measure of depression consistent with Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria. The self-report rating scale is 0-3 for each symptom, with higher scores indicating greater symptom severity. PHQ-9 has demonstrated good psychometric properties including criterion, construct, and external validity, and sensitivity (88%) and specificity (88%) for major depressive disorder.
Change in Quality of Life Measured by WHOQOL-BREF: Social Relationships and Environment Scales | Months 0 (baseline), 3, 6, and 12
  The self-report 26-item WHOQOL-BREF was multi-nationally developed to assess QOL related to physical health, psychological well-being, social relationships, and environment. The Social Relationships scale assesses facets of quality of life related to personal relationships, social support, and sexual activity. The Environment scale assesses facets related to quality of life including physical safety and security, accessibility and quality of health and social care, and participation in social and leisure opportunities.
Patient Satisfaction Measured By Satisfaction with Therapy and Therapist Scale-Revised (STTS-R) | Months 3, 6, and 12
  The 13-item self-report STTS-R comprises two scales (Satisfaction with Therapy and Satisfaction with Therapist), both with documented reliability and validity.
Assessing Treatment Dropout Measured by Completion of Less than 8 Sessions | Across intervention
  Treatment dropout is defined as completion of < 8 sessions, corresponding to the median effective dose. The number of sessions completed will be identified through mandatory session notes completed by clinicians for each study visit.

OTHER OUTCOMES:
Minority Stress Measured by Cultural Assessment of Risk for Suicide (CARS) Minority Stress Subscale - Moderator | Months 0 (baseline), 3, 6, and 12
  The adapted minority stress subscales of the CARS have been established as a measure of general minority stress. This subscale consists of five items answered on a 6-point scale ranging from "strongly disagree" to "strongly agree."
Substance Use Measured Alcohol and Substance, Smoking, and Substance Involvement Screening Test (ASSIST) - Moderator | Months 0 (baseline), 3, 6, and 12
  The ASSIST is a self-report measure of substance use that gives a score ranging from 0-39, with higher scores reflecting greater substance use involvement, and validated cutoff scores for low, moderate, or high risk substance use involvement.

CONTACTS AND LOCATIONS:
Overall Officials: Annesa P Flentje, PhD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University, Palo Alto, California
  - UCSF Alliance Health Project, San Francisco, California

IPD SHARING:
Plan to Share IPD: No
Individual participant data will only be available to the researchers affiliated with this clinical trial. All data are de-identified and stored on a firewall-protected server.